CLINICAL TRIAL: NCT05220878
Title: Multicenter Randomized Double-blind Comparative Study of Clinical Efficacy and Safety of GNR-069 (JSC "GENERIUM", Russia) and Nplate (Amgen Europe BV, The Netherlands) in Patients With Idiopathic Thrombocytopenic Purpura
Brief Title: Comparative Study of Clinical Efficacy and Safety of GNR-069 and Nplate in Patients With ITP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RMP-ITP-III; № 407 eff. date 29 July 2021 (Other: Ministry of Health of the Russian Federation)
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: Idiopathic thrombocytopenic purpura; ITP; Thrombocytopenia; Thrombocytopoiesis; Bleeding; Hemorrhagic syndrome; Petechial rash; Ecchymosis; Fc-peptide; Recombinant DNA technology; Thrombopoietin receptors; Platelet formation; Fc fragment of human immunoglobulin IgG 1; Low platelet count; ITP treatment; Platelets; Haemorrhage; Platelet destruction; Impaired thrombopoiesis; Megakaryocytes; Autoantibodies; Splenectomy; Cytotoxic; T cells; Thrombopoietin receptor agonists; TPO-RAs; romiplostim; Nplate
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia; Hemorrhage; Purpura; Ecchymosis | interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNR-069 (Experimental): Main group (80 patients) - multiple weekly subcutaneous injections of GNR-069, doses are calculated individually.
  Interventions: Biological: GNR-069
- Nplate (Active Comparator): Control group (80 patients) - multiple weekly subcutaneous injections of Nplate, doses are calculated individually.
  Interventions: Biological: Nplate

INTERVENTIONS:
Biological: GNR-069 — Once a week as a subcutaneous injection. The initial dose is 1 mcg/kg.
  Other Names: romiplostim
  Arms: GNR-069
Biological: Nplate — Once a week as a subcutaneous injection. The initial dose is 1 mcg/kg.
  Other Names: romiplostim
  Arms: Nplate

SUMMARY:
It is a phase III multicenter randomized double-blinded comparative study of clinical efficacy and safety of GNR-069 and Nplate in patients with idiopathic thrombocytopenic purpura

DETAILED DESCRIPTION:
The drug GNR-069(JSC "GENERIUM", Russia) is biosimilar to the original drug Nplate. This study is aimed to compare the clinical efficacy and safety of the drug GNR-069 and the drug Nplate to register of the drug GNR-069 in the Russian Federation for therapy in patients with idiopathic thrombocytopenic purpura (ITP). The study also provides for the evaluation of pharmacokinetic parameters and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent Form to participate in the study;
2. Men and women aged 18-75 years inclusive at the time of signing the Informed Consent Form;
3. Documented diagnosis of ITP with a disease duration of more than 12 months from the moment of confirmation of the diagnosis by bone marrow aspirate or biopsy results;
4. A. For patients who have not had splenectomy:

   * established absence/loss of response to therapy with at least one drug of fist-line treatment for ITP (which include GCs an IVIG); OR
   * the occurrence of side effects during the course of therapy with the drug of the fist-line, making it impossible to use it further;

   B. For patients who underwent splenectomy:

   • loss/lack of response to splenectomy;
5. Thrombocytopenia ≥30.0 x 109/L - <50.0 x 109/L with severe hemorrhagic syndrome or thrombocytopenia <30.0 x 109/l, regardless of the presence of hemorrhagic syndrome, according to the results of platelet count conducted in a local laboratory for 7 days before the start of therapy with investigational or reference drug;
6. Patients receiving GCs, azathioprine and danazole should receive these drugs in a maintenance dose for at least 4 weeks before starting therapy with investigational or reference drug;
7. Consent of study participants with preserved childbearing function to use reliable methods of contraception (a combination of at least two methods, including 1 barrier method, for example, the use of a condom and spermicide) from the moment of signing the Informed Consent Form and 3 months after the last administration of investigational or reference drug.

Exclusion Criteria:

1. Hypersensitivity to the components of investigational or reference drug or E. coli proteins ;
2. Unresolved severe hemorrhagic syndrome requiring emergency treatment at the time of initiation of study or reference drug therapy ;
3. Fisher-Evans Syndrome;
4. Conditions with a high risk of thromboembolic complications ;
5. Myelodysplastic syndrome and/or bone marrow transplantation in anamnesis;
6. Deviations of clinical and laboratory parameters according to the results of studies of blood samples taken during the screening period;
7. Positive test results for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV);
8. Pregnancy or breastfeeding;
9. Use of drugs:

   * romiplostim used less than 3 weeks before treatment with study or reference drug;
   * IVIG - less than 2 weeks prior to initiation of study or reference drug therapy;
   * eltrombopag - used less than 2 weeks before treatment with study or reference drug, or planned to use eltrombopag while the patient is participating in this study;
   * rituximab - used less than 14 weeks before treatment with study or reference drug, or planned to use rituximab while the patient is enrolled in this study;
   * cyclophosphamide, cyclosporine, vincristine, vinblastine and other drugs used to treat ITP not listed above and not included in the list of drugs approved for use during the study - use less than 8 weeks before the start of therapy with the study or reference drug or the use of any of these drugs is planned during the patient's participation in this study;
   * preparations of any hematopoietic growth factors - use less than 8 weeks before the start of therapy with an investigational or reference drug;
   * Influenza vaccines - less than 21 days prior to start of treatment with study or reference drug;
   * vaccines to prevent novel coronavirus disease (COVID-19) - completion of the vaccination program less than 21 days prior to the start of study or reference drug therapy;
   * other vaccines - less than 8 weeks prior to start of treatment with study or reference drug;
10. Splenectomy within 12 weeks prior to screening;
11. Participation in any clinical trials and/or use of unregistered drugs within 4 weeks prior to screening or 5 drug half-lives (whichever is greater);
12. Any other disease or condition that, in the opinion of the investigator, may preclude the patient from participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving sustained response to treatment | 26 weeks
  A sustained response to treatment is defined as the number of platelets ≥ 50.0 x 109/L for at least 9 out of 12 consecutive visits during the treatment period with the study or reference drug.

SECONDARY OUTCOMES:
Proportion of patients who achieve stable platelet count during treatment with investigational or reference drug | 26 weeks
  Stable platelet count is defined as the number of platelets ≥ 50.0 x 109/L for at least 4 consecutive weeks without dose adjustment.
Time from initiation of therapy with investigational or reference drug to reaching a stable platelet count | 26 weeks
Number of cases of emergency therapy for severe hemorrhagic syndrome during the treatment period, starting from the second week of therapy with the investigational or reference drug | 25 weeks
Number of clinically significant bleeding episodes during the treatment period, starting from the second week of therapy with investigational or reference drug | 26 weeks
  Bleeding episode ≥ Grade 2 according to CTCAE version 5.0 is considered clinically significant
Change in ITP-specific bleeding assessment tool (ITP-BAT) scores at last visit from baseline at screening | 26 weeks
Proportion of patients with no/loss of response to treatment with investigational or reference drug | 26 weeks
Proportion of patients receiving approved ITP prophylactic drugs (glucocorticosteroids, azathioprine, danazol) in this study at the time of randomization | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, MSc, Study Chair — AO GENERIUM
Locations (18):
- Russia (18):
  - Federal State Budgetary Educational Institution of Higher Education "Bashkir State Medical University" of the Ministry of Health of the Russian Federation, Ufa, Bashkortostan Republic
  - State Budgetary Institution of Healthcare Irkutsk awarded the "Sign of Honor" Order Regional Clinical Hospital, Irkutsk, Irkutsk Oblast
  - State Budgetary Health Institution of the Kaluga Region "Kaluga Regional Clinical Hospital", Kaluga, Kaluga Oblast
  - State Autonomous Healthcare Institution "Kuzbass Clinical Hospital named after S.V. Belyaev", Kemerovo, Kemerovo Oblast
  - State budgetary institution of health care of the Nizhny Novgorod region "Nizhny Novgorod Regional Clinical Hospital named after N. A. Semashko", Nizhny Novgorod, Nizhny Novgorod Oblast
  - Llc "Medis", Nizhny Novgorod, Nizhny Novgorod Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Novosibirsk State Medical University" of the Ministry of Health of the Russian Federation, Novosibirsk, Novosibirsk Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Rostov State Medical University" of the Ministry of Health of the Russian Federation, Rostov-on-Don, Rostov Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Samara State Medical University" of the Ministry of Health of the Russian Federation, Samara, Samara Oblast
  - Federal State Budgetary Educational Institution of Higher Education "Saratov State Medical University named after V.I. Razumovsky" of the Ministry of Health of the Russian Federation, Saratov, Saratov Oblast
  - State Health Institution of the Tula Region "Tula Regional Clinical Hospital", Tula, Tula Oblast
  - State Budgetary Institution of Healthcare of the city of Moscow "Moscow Clinical Scientific and Practical Center named after A.S. Loginov" Department of Health of the city of Moscow., Moscow
  - Federal State Budgetary Institution "National Medical Research Center for Hematology" of the Ministry of Health of the Russian Federation, Moscow
  - State budgetary health care institution of the city of Moscow "Clinical Hospital named after S.P. Botkin" of the Department of Health of the city of Moscow, Moscow
  - State budgetary health care institution of the city of Moscow "City Clinical Hospital named after V.V. Veresaev of the Department of Health of the City of Moscow", Moscow
  - State Budgetary Health Institution of the Moscow Region "Moscow Regional Research Clinical Institute named after M.F. Vladimirsky", Moscow
  - Federal State Budgetary Institution "National Medical Research Center named after V.A. Almazov" of the Ministry of Health of the Russian Federation, Saint Petersburg
  - Municipal budgetary institution "Central City Hospital No. 7", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No